CLINICAL TRIAL: NCT05085197
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Single-ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of STSA-1005 Following Intravenous Infusion in Healthy Subjects
Brief Title: The Safety and Tolerability of STSA-1005 Following Intravenous Infusion in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSA-1005-01
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2021-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1:1mg/kg (Experimental): All participants (fasted) received either 1mg/kg of STSA-1005 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1005 injection; Drug: Placebo
- Cohort 2:2.5mg/kg (Experimental): All participants (fasted) received either 2.5mg/kg of STSA-1005 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1005 injection; Drug: Placebo
- Cohort 3:5mg/kg (Experimental): All participants (fasted) received either 5 mg/kg of STSA-1005 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1005 injection; Drug: Placebo
- Cohort 4:10mg/kg (Experimental): All participants (fasted) received either 10 mg/kg of STSA-1005 as a single dose or dose-matched placebo.
  Interventions: Drug: STSA-1005 injection; Drug: Placebo

INTERVENTIONS:
Drug: STSA-1005 injection — Intravenous injection
  Arms: Cohort 1:1mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 1:1mg/kg
Drug: STSA-1005 injection — Intravenous injection
  Arms: Cohort 2:2.5mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 2:2.5mg/kg
Drug: STSA-1005 injection — Intravenous injection
  Arms: Cohort 3:5mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 3:5mg/kg
Drug: STSA-1005 injection — Intravenous injection
  Arms: Cohort 4:10mg/kg
Drug: Placebo — Intravenous injection
  Arms: Cohort 4:10mg/kg

SUMMARY:
This was a single ascending dose, randomized, double-blind study assessing the safety, tolerability and pharmacokinetics of STSA-1005 in healthy participants. Four kinds different doses and dose-matched placebo were administered under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are able to understand and are willing to sign the informed consent form (ICF).
2. Subjects (male or female) must be ≥18 to ≤65years of age inclusive.
3. Healthy subjects according to the results of medical history, physical examination, vital signs, ECG, and clinical laboratory examination. The Investigator considers that the subjects are in good health with no clinically significant heart, liver, kidney, digestive tract, nervous system, respiratory system, mental disorders, and metabolic disorders.
4. Subjects with a body mass index (BMI) of 20-32kg/m^2, inclusive.
5. (1)If a subject is a female of childbearing potential - she should agree to use one of the accepted contraceptive regimens from at least 30 days before screening, during the study, and for at least 3 months after administration of the study treatment.1)An acceptable method of contraception includes one of the following:

   * Abstinence from heterosexual intercourse;

     * Hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch);

       * Intrauterine device (with or without hormones). 2)OR she should agree to use a double-barrier method (e.g., condom and spermicide) during the study and for at least 3 months after administration of the study treatment.

         (2)If a subject is a female of non-childbearing potential - she should be surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or in a menopausal state (at least 1 year without menses), as confirmed by Follicle stimulating hormone (FSH) levels (≥40 mIU/mL).
6. A male study subject that engages in sexual activity that has the risk of pregnancy must agree to use a double-barrier method (e.g., condom and spermicide) and agree to not donate sperm during the study and for at least 90 days after administration of the study treatment.
7. Subjects understand the risks of the study, can comply with the study protocol, and complete the study.

Exclusion Criteria:

1. History of cardiovascular, respiratory, kidney, liver, metabolic, endocrine, gastrointestinal, blood, neurological, skin, psychiatric, cancer, or other major serious diseases that in the judgment of the Investigator might put the subject at risk on this study.
2. History of tuberculosis (active or latent) irrespective of treatment status or infection within the past 4 weeks or history of recurrent infections.
3. History of or current active autoimmune disease or immunodeficiency disease.
4. Subjects who have a history of clinically significant drug allergy or atopic allergic disease or known allergic reaction or hypersensitivity to the study treatment or its excipients according to the judgment of the Investigator.
5. Subjects who have a history of drug abuse in the 12 months before screening or who have a positive urine drug tests at the time of screening.
6. Subjects who have taken biologic agents within 3 months or 5 times the half-life (whichever is longer) before screening, or who have taken drugs that may affect immune function within 6 months or 5 times the half-life (whichever is longer) before screening, or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homoeopathic preparations, vitamins, and minerals) within 7 days prior to IMP administration.
7. Subjects who have received treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to screening or 90 days for biologic compounds prior to screening.
8. Blood donation (excluding plasma donation) of approximately 500 mL within 56days before screening or plasma donation within 7 days before screening.
9. Those whose daily consumption of alcohol at the time of screening or at any time within the prior 6 months is more than 2 standard drinks, where 1 standard drink = 355 mL or 12 oz (1can) of regular-strength (5%) beer; 150 mL or 5 oz wine; 45 mL or 1.5 oz liquor/spirits (40%) or who are positive for alcohol tests during the screening period.
10. Female subjects who are breastfeeding or pregnant or who have positive serum pregnancy test during the screening period and on admission.
11. Subjects who have difficulty in venous blood collection or who exhibits risk of fainting after blood collections or with the site of needles.
12. Human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody test results are positive during the screening period.
13. Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.
14. Subjects who have participated in any vaccine clinical study as subjects within 3 months before enrollment or plan to receive live vaccines during the study period, and subjects who have received inactivated vaccines 28 days prior to the IMP administration or plan to receive inactivated vaccines within 2 months after the end of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Serious Adverse Events, Clinically Significant Laboratory Abnormalities, Electrocardiogram Abnormalities, Vital Signs Abnormalities and Physical Examination Abnormalities. | Day 1 through Day 57

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to 1344 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1005 in healthy adult subjects
Area under the plasma concentration-time curve from time 0 to the collection time point t of the last measurable concentration (AUC0-t) | Up to 1344 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1005 in healthy adult subjects
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-∞) | Up to 1344 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1005 in healthy adult subjects
Time of maximum concentration (Tmax) | Up to 1344 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1005 in healthy adult subjects
Elimination half-life (t1/2) | Up to 1344 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1005 in healthy adult subjects
Fraction of drug eliminated per unit of time (Kel) | Up to 1344 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1005 in healthy adult subjects
Last measurable concentration (Clast) | Up to 1344 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1005 in healthy adult subjects
Mean residence time (MRT) | Up to 1344 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1005 in healthy adult subjects
Clearance (CL) | Up to 1344 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1005 in healthy adult subjects
Apparent volume of distribution (Vz/F) | Up to 1344 hours postdose
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1005 in healthy adult subjects
The number of subjects with anti-drug antibody (ADA) and neutralizing antibody (NAb) | Up to 1344 hours postdose
Change from baseline in numbers of neutrophils and monocytes | Up to 1344 hours postdose
Changes of granulocyte macrophage colony-stimulating factor (GM-CSF) receptor occupancy (RO) after the administration compared with the baseline | Up to 1344 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- AltaSciences Clinical Kansas, Inc, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No